CLINICAL TRIAL: NCT03921905
Title: Peripheral Artery Disease in Patients With Stable Coronary Artery Disease in General Practice: Prevalence, Management and Clinical Outcomes.
Acronym: PAD&CAD
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IRFMN-7825
Record Dates: First submitted 2019-04-01; First posted 2019-04-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Coronary Artery Disease; General Practice; Ankle-brachial index (ABI)
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CAD: In this study will be included patients with stable CAD
  Interventions: Diagnostic Test: ABI measurement

INTERVENTIONS:
Diagnostic Test: ABI measurement — ABI measurement wil be done with an automatic device to diagnose PAD in patients with CAD

SUMMARY:
Patients with lower extremity peripheral artery disease (PAD) are at risk of developing major adverse limb events and have a similar cardiovascular (CV) morbidity and mortality to those with coronary artery disease (CAD) with which is associated in most cases with a more severe prognosis. Because of higher risk conferred by concomitant PAD an early diagnosis is recommended in subjects with CAD. PAD can be diagnosed relatively easily and noninvasively with the ankle-brachial index (ABI) measure. An ABI ≤0.9 is an indicator of the presence of lower extremity PAD, indicating athero-occlusive arterial disease while >1.3/1.4 indicates an incompressible ankle arteries. However, ABI is not routinely applied in the clinical practice. Data on prevalence of PAD are scanty and in patients with stable CAD are lacking. The under-diagnosis of PAD may be a barrier to the use of treatments to improve prognosis. The primary aim of this study is to assess the coexistence of PAD in subjects with stable CAD and to evaluate the management and the prognosis of these patients in primary care at 12-month after the inclusion in the study.

DETAILED DESCRIPTION:
National, multicentre, observational, prospective study. This study will be carried out with the collaboration with Study Center for Primary Care and with the Italian Society of Angiology and Vascular Medicine (SIAPAV).

The eligible patients with stable CAD will be called by General Practitioners (GPs).

For all patients who agree to participate in the study and sign the consent, two visits will be done at baseline and after 12 months.

At baseline will be collected information on socio-demographic and anthropometric data, blood pressure, heart rate, CV risk factors, medical history, lifestyle habits, PAD stage (for patient with abnormal ABI) and pharmacological therapy. ABI measurement will be done using an automatic simple device. In case of abnormal ABI value, a SIAPAV vascular specialist, at GP's office, will confirm it using the standard manual continuous wave (CW) Doppler.

At follow-up visit the following information will be collected the: referral to vascular specialist (if requested, at discretion of the GP), relevant change in pharmacological therapy, major CV events and progression of PAD, limb and coronary artery revascularizations, amputations, major bleeding, and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a diagnosis of stable CAD as follows: acute myocardial infarction or percutaneous coronary revascularization or coronary artery bypass graft surgery occured at least 12 months before entering the study or chronic stable angina.

Exclusion Criteria:

* Mental illness limiting the capacity of self-care or any condition limiting seriously the life expectancy less than 12 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of stable CAD in charge of GPs, giving the consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
To know the prevalence of PAD in patients with CAD using the automatic device MESI ankle-brachial pressure index (ABPI) MD® | 1 day
  The prevalence of PAD will be diagnosed measuring the ankle-brachial-index (ABI) determined by dividing the higher systolic pressure measured at the ankle of both legs by the brachial arterial systolic pressure. An ABI value <=0.9 is an indicator of the presence of PAD indicating athero-occlusive arterial disease while >1.3/1.4 indicates an incompressible ankle arteries. The ABI measurement will be performed using the automatic device MESI ABPI MD.

SECONDARY OUTCOMES:
To measure the Blood pressure (mmHg) | 1 day
To measure the Heart rate (bpm) | 1 day
To measure the Weight (kg) | 1 day
To measure the Height (cm) | 1 day
To measure the Body mass index (Kg/m2) | 1 day
To measure the Ankle Brachial Index (ABI) Value | 1 day
Clinical History of Limb peripheral artery revascularization | 1 day
Clinical History of Limb or foot amputation for arterial vascular disease | 1 day
Clinical History of Clinical presentation of lower extremity disease | 1 day
Clinical History of Aortic aneurysm | 1 day
Clinical History of Carotid artery stenosis | 1 day
Clinical History of Heart Failure | 1 day
Clinical History of Atrial Fibrillation or Flutter | 1 day
Clinical History of Hypertension | 1 day
Clinical History of Dyslipidemia | 1 day
Clinical History of Chronic Kidney disease | 1 day
Clinical History of Stroke | 1 day
Clinical History of Transient ischemic attack | 1 day
Clinical History of Bleeding | 1 day
Clinical History of cancer | 1 day
The dietary habits | 1 day
  The Mediterranean Diet Questionnaire (Prevention with a Mediterranean Diet PREDIMED -14 Items) will be administered
Physical activity | 1 day
  The Physical activity Questionnaire (BRFSS 2 items) will be administered
Total cholesterol (mg/dL) | 1 day
LDL cholesterol (mg/dL) | 1 day
HDL cholesterol (mg/dL) | 1 day
Triglycerides (mg/dL) | 1 day
Glycemia (mg/dL) | 1 day
Glycated hemoglobin (only for patients with diabetes mellitus) (%) | 1 day
Creatinine (mg/dL) | 1 day
Alanine aminotransferase (ALT) (U/L) | 1 day
Aspartate aminotransferase (AST) (U/L) | 1 day
Hemoglobin (g/dL) | 1 day
Platelet count (x 103μL) | 1 day
Hematocrit (%) | 1 day
Red blood cells (x10^3 ml) | 1 day
White blood cells (x10^3 ml) | 1 day
Marital status | 1 day
Education Status | 1 day
Employment status | 1 day

OTHER OUTCOMES:
The incidence of Acute coronary syndrome | 12 months
The incidence of Stroke | 12 months
The incidence of Transient ischemic attack | 12 months
The incidence of Heart Failure | 12 months
The incidence of Atrial fibrillation or Flutter | 12 months
The incidence of Coronary artery revascularization | 12 months
The incidence of Hospitalization for worsening of PAD | 12 months
The incidence of Limb peripheral artery revascularization | 12 months
The incidence of Lower limb amputation for arterial vascular disease | 12 months
The incidence of Major bleeding (bleeding leading to hospitalization, bleeding requiring surgical procedures to manage the bleeding, bleeding requiring blood trabsfusion) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marta Baviera, PharmD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (4):
- Italy (4):
  - MEDICOOP Genova, Genova, GE
  - Cooperativa Medici Milano Centro, Milan, MI
  - MEDICOOP S. Agata, Reggio Calabria, RC
  - ROMAMED Service, Rome, RM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Baviera M, Foresta A, Fernandez LO, Torrigiani G, Tettamanti M, Roncaglioni MC, Cimminiello C; PAD, C. A. D. Study Group. Peripheral artery disease in patients with stable coronary artery disease in general practice: results from an Italian nationwide study-PAD & CAD study. Intern Emerg Med. 2025 Jan;20(1):159-169. doi: 10.1007/s11739-024-03771-9. Epub 2024 Sep 30. PMID 39347889